CLINICAL TRIAL: NCT05641376
Title: Nebulized Versus Intravenous Dexmedetomidine for Managing Sevoflurane Induced Emergence Agitation After Pediatric Tonsillectomy
Brief Title: Nebulized Versus Intravenous Dexmedetomidine for Sevoflurane Induced Emergence Agitation After Pediatric Tonsillectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Aboulfotouh Mohammed, lecturer of Anesthesia and icu, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 60757593
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nebulized Dexmedetomidine (Active Comparator): Children will receive a nebulized dexmedetomidine 2 mic/ kg diluted in 3 ml of 0.9% saline 1 h before induction of anaesthesia.
  Interventions: Drug: Nebulized Dexmedetomidine
- Intravenous Dexmedetomidine (Active Comparator): Children will receive intravenous (IV) dexmedetomidine 1mic/kg diluted in 10 ml of 0.9% saline over 10 minutes after anesthesia induction.
  Interventions: Drug: Intravenous Dexmedetomidine

INTERVENTIONS:
Drug: Nebulized Dexmedetomidine — Children will receive a nebulized dexmedetomidine 2 mic/ kg diluted in 3 ml of 0.9% saline 1 h before induction of anaesthesia by standard hospital jet nebulizer via a mouthpiece with a continuous flow of 100% oxygen at 6 L /min for 10-15 min. Treatment will be stopped when the nebulizer began to sputter. At end of nebulizer administration, they will be observed for 30 min before induction of general anaesthesia. then the children will be transferred to the operation room and will receive intravenous (IV) normal saline 0.9% in 10 ml volume over 10 minutes after anesthesia induction.
  Arms: Nebulized Dexmedetomidine
Drug: Intravenous Dexmedetomidine — Children will receive nebulized 3 ml of 0.9% normal saline 1 h before induction of anaesthesia by standard hospital jet nebulizer via a mouthpiece with a continuous flow of 100% oxygen at 6 L /min for 10-15 min. then the children will be transferred to the operation room and will receive intravenous (IV) dexmedetomidine 1mic/kg diluted in 10 ml of 0.9% saline over 10 minutes after anesthesia induction.
  Arms: Intravenous Dexmedetomidine

SUMMARY:
Pediatric patients undergoing tonsillectomy and adenoidectomy usually have a high incidence of postoperative EA, which increases the risk of developing postoperative airway obstruction and respiratory depression due to anatomical characteristics of operative location and increased susceptibility to opioid analgesics. the study will compare between nebulized and intravenous bolus of dexmedetomidine as a prophylaxis against postanesthetic emergence agitation in children undergoing tonsillectomy, adenoidectomy or adeno-tonsillectomy procedures.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* Children scheduled for tonsillectomy with or without adenoidectomy with or without myringotomy, and/or tympanostomy tube insertion.

Exclusion Criteria:

* Patient's guardian refusal to participate in the study.
* Children with Behavioral changes; physical or developmental delay; neurological disorder or psychological disorder.
* Children on sedative or anticonvulsant medication.
* history of sleep apnea
* significant organ dysfunction, cardiac dysrhythmia, congenital heart disease
* Known allergy to the study drugs.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative Emergence agitation will be evaluated using the Paediatric Anaesthesia Emergence Delirium scale | 60 minutes
  Paediatric Anaesthesia Emergence Delirium (PAED) scale will be used to evaluate emergence agitation upon admission to the PACU (0 min, baseline) and at 5, 10, 20, 30, 45, and 60 min until discharge from the PACU. The highest EA scores observed during this period will be recorded.
  PAED score ≥ 10 will be considered to be a diagnostic endpoint for the development of agitation.

SECONDARY OUTCOMES:
Postoperative pain | 60 minutes
  Postoperative pain will be recorded using FLACC scale at 5, 10, 20, 30, 45, and 60 min until discharge from the PACU.
emergence agitation (EA) onset | 60 minutes
  Emergence agitation onset time was defined as the interval from the extubation to the occurrence.
Emergence Agitation duration | 60 minutes
  Emergence agitation duration was the time from Emergence agitation onset to its cessation

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt